CLINICAL TRIAL: NCT04537936
Title: Adaptation and Pilot Feasibility of a Psychotherapy Intervention for Latinos With Advanced Cancer
Brief Title: Psychotherapy Intervention for Latinos With Adv Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Lincoln Medical and Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-076A(20)
Record Dates: First submitted 2020-09-01; First posted 2020-09-03 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor; Solid Tumor, Adult; Solid Tumor, Unspecified, Adult
Keywords: Stage III solid tumor cancer; Stage IV solid tumor cancer; Stage III cancer; Stage IV cancer; Spanish; Memorial Sloan Kettering Cancer Center; 15-076
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meaning Centered Psychotherapy for Latinos (MCP-L) (Experimental)
  Interventions: Behavioral: Meaning Centered Psychotherapy for Latinos; Behavioral: Functional Assessment of Cancer Therapy - Spiritual Well-Being Scale; Behavioral: Meaning Centered Psychotherapy for Latinos for Waitlist Control Patients; Behavioral: Pre-assessment questionnaire
- Control (Active Comparator)
  Interventions: Behavioral: Meaning Centered Psychotherapy for Latinos; Behavioral: Functional Assessment of Cancer Therapy - Spiritual Well-Being Scale; Behavioral: Meaning Centered Psychotherapy for Latinos for Waitlist Control Patients; Behavioral: Pre-assessment questionnaire

INTERVENTIONS:
Behavioral: Meaning Centered Psychotherapy for Latinos — MCP-L consists of seven-60 minute-individual sessions. The seven sessions are expected to be delivered every week or every two weeks over a span of 7-14 weeks.
  Other Names: MCP-L
Behavioral: Functional Assessment of Cancer Therapy - Spiritual Well-Being Scale — Determines the degree of spiritual well-being
Behavioral: Meaning Centered Psychotherapy for Latinos for Waitlist Control Patients — Waitlist Control Patients in the control condition will be allocated to a waitlist group to receive the intervention approximately three months after randomization.
Behavioral: Pre-assessment questionnaire — Which includes 10 standardized scales Assessment/Evaluation Plan, Phase 1, 4 - Quantitative Measure Questionnaire).The interview guide will inquire about the comprehension and acceptability of, and alternative options for, these intervention components.

SUMMARY:
The purpose of this study is to adapt a counseling intervention called Meaning Centered Psychotherapy to make it culturally relevant for Latinos. Cancer affects patients and their loved ones. Latinos often experience greater challenges due to the cancer. However, few studies and interventions focus on Latinos. We are interested in understanding what affects Latino patients' quality of life, and how to improve it

DETAILED DESCRIPTION:
Overview of the Study. This project has 5 phases. In phases 1 and 2 the study team will work to gain an understanding of the sources of meaning, hope, legacy and identity in Latino patients with advanced cancer; and to explore the acceptability and feasibility of applying IMCP to Latinos diagnosed with advanced cancer. A convergent mixed-methods design will be utilized with a sample of 200 Latino patients diagnosed with advanced cancer for the quantitative phase, and a nested cohort of 14-20 for the qualitative phase from two cancer centers in New York City: Memorial Sloan Kettering Cancer Center (MSKCC) and Lincoln Medical and Mental Health Center (LMC), a public hospital localized in a Latino-dense region. We will also recruit eligible cancer patients serviced through Dr. Gany's Integrated Cancer Care Access Network (ICCAN). The Integrated Cancer Care Access Network (ICCAN) of MSKCC's Immigrant Health and Cancer Disparities Service (IHCD) enrolls patients at eleven hospital-based cancer clinics in New York City with large numbers of immigrant and low-income patients. ICCAN uses bilingual Access Facilitators to assist patients in accessing and utilizing health, social, and financial services. Identified needs of the patients, range from psychosocial support, to health literacy, child care, financial, housing and legal concerns. Patients enrolled to the ICCAN program are actively obtaining support from Access Facilitators throughout their treatment period. Access Facilitator will refer eligible patients to the study team for recruitment.

Before moving to phase 3, we will adapt and transcreate (the source text is rewritten to convey the concepts and achieve the aims of the source text, while accounting for both language and cultural considerations) the manual based on the phase 1 and 2 findings. In the phase 3 (Key Informant feedback), mental health providers will be interviewed to explore additional needed adaptations.

Phase 4 will consist of pre-piloting or interviewing patients to assess the comprehension and acceptability of the adapted intervention. Patient Feedback phase, key components of the intervention will be pre-piloted with 6-10 patients across MSKCC and, Lincoln Medical and Mental Health Center (LMC)

Participants who express concerns or request assistance related to COVID-19 will be referred to publicly available resources as needed (e.g., call 311 for access to health care or food panties, etc.) and will be noted in internal tracking logs.

Phase 5 Randomized Controlled Pilot Study Phase will collect preliminary data on the feasibility of recruitment, retention and adherence and acceptability of content of Meaning-Centered Psychotherapy for Latinos (MCP-L) and key outcomes (spiritual well-being, depression, anxiety, hopelessness, and quality of life). Additional information will be collected, specifically scales measuring , attitudinal familism, acculturation, fatalism, religiosity, literacy , and racial microaggressions which will inform the design of a future large-scale randomized clinical trial of the culturally adapted intervention. A sample of 60 Spanish-speaking advanced cancer patients will be enrolled and randomized evenly to MCP-L or to Enhanced Usual Care (EUC) control.

Eligible patients for Phase 5 will meet the same criteria as Phase 1 patients ; however patients who score > 4 on the Distress Thermometer will be recruited to Phase 5, and patients who score < 4 will be recruited to Phase 1.

ELIGIBILITY:
Inclusion Criteria:

Phase I: Quantitative

* Diagnosed with stages III or IV solid tumor cancer *(as per self report for ICCAN patients)
* Age 18 or older
* As per self report, Latino/a or Hispanic ethnicity
* As per self report, fluent in oral Spanish (monolingual) or fluent in oral Spanish and English (bilingual)

Phase 2: Qualitative

* Enrolled in the quantitative phase of study (as seen above)
* Completes the quantitative phase questionnaire
* Scores above or below the threshold for the Distress Thermometer (DT≥4 or ≤3)
* In the judgment of the investigator, willing and able to be interviewed in Spanish only
* Agrees to be audio- recorded

Phase 3: Provider Feedback

* Professionals working in the mental health field;
* Have a caseload of five or more Latino cancer patients per month
* Able to communicate and read in Spanish
* Agrees to be audio or video-recorded

Phase 4: Patient Feedback

* Diagnosed with stages III or IV solid tumor cancer *(as per self report for ICCAN patients)
* Age 18 or older
* As per self report, Latino/a or Hispanic ethnicity
* In the judgment of the investigator, willing and able to be interviewed in Spanish only
* Agrees to be audio-recorded

Phase 5: Pilot RCT

* Diagnosed with stages III or IV solid tumor cancer
* Age 18 or older
* Latino/a or Hispanic ethnicity
* Fluent in oral Spanish (monolingual or bilingual)
* Scores above the threshold for the Distress Thermometer (DT≥4)
* Agrees to be audio-recorded

Exclusion Criteria:

Phase 1: Quantitative

* In the judgment of the treating physician and/or the consenting professional, presence of significant cognitive impairment (i.e., delirium or dementia) sufficient to preclude meaningful informed consent and/or data collection
* In the judgment of the consenting professional, significant or major disabling medical or psychiatric condition sufficient to preclude meaningful informed consent, interview, or completion of assessment measures (patients whose psychiatric disorder is well controlled by treatment will be eligible)

Phase 2: Qualitative

* In the judgment of the treating physician and/or the consenting professional, presence of significant cognitive impairment (i.e., delirium or dementia) sufficient to preclude meaningful informed consent and/or data collection
* In the judgment of the consenting professional, significant or major disabling medical or psychiatric condition sufficient to preclude meaningful informed consent, interview, or completion of assessment measures (patients whose psychiatric disorder is well controlled by treatment will be eligible)

Phase 4: Patient Feedback

* Diagnosed with a major disabling medical or psychiatric condition
* Unable to understand the consent procedure
* Too ill to participate, all as reported by the patient and/or determined by the investigator's judgment.

Phase 5: Pilot RCT

* Diagnosed with a major disabling medical
* Diagnosed with a major disabling psychiatric condition
* Unable to understand the consent procedure
* Too ill to participate, all as reported by the patient and/or determined by the investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Spiritual Well-Being measured with the FACIT Spiritual Well-Being Scale | Change from baseline to post assessment 7-14 weeks after
  FACIT Spiritual Well-Being Scale is a brief self-report measure designed to assess the nature and extent of individual spiritual well-being. This measure, which generates two sub-scales, one corresponding to Faith (the importance of faith and spirituality) and a second assessing Meaning-Peace (one sense of meaning and purpose in life), has been demonstrated to have strong internal reliability for both the total score as well as each subscale (coefficient alpha equals .87 for the total scale, .88 for the faith factor and .81 for the meaning factor). In additional, strong support for the external validity of this measure has been demonstrated in a several large samples of cancer and AIDS patients and with Spanish speaking populations.

SECONDARY OUTCOMES:
Depression and Anxiety measured with the Hospital Anxiety and Depression Scale | Change from baseline to post assessment 7-14 weeks after
  The Hospital Anxiety and Depression Scale (HADS) is a validated scale used to measure anxiety and depression. This scale has been validated against structured or semi-structured clinical interviews, the gold standard for the assessment of mental disorders, in a significant number of studies. Further strengths of this scale for the assessment of emotional distress in cancer patients stem from the joint assessment of anxiety and depressive symptoms without referring to physical symptoms of anxiety or depression. Given the high comorbidity of anxiety of cancer as well as the systematic exclusion of confounding physical symptoms, the scale seems especially appropriate for use in this patient group. The HADS consists of 14 items which reflect a 7-item anxiety and a 7-item depression subscale. This scale has sound psychometric properties in Spanish.
Hopelessness measured with the Beck Hopelessness Scale | Change from baseline to post assessment 7-14 weeks after
  The Beck Hopelessness Scale (BHS) comprises 20 true/false questions that assess degree of pessimism and hopelessness. Several studies have demonstrated a high degree of internal consistency and construct validity. Scores ranging from 4 to 8 typically indicate a "mild" degree of hopelessness, 9 to 12 correspond to "moderate" hopelessness, and scores about 12 reflect "severe" levels of hopelessness.
Quality of life measured with the FACIT Spiritual Well-Being Scale | Change from baseline to post assessment 7-14 weeks after
  The FACIT Spiritual Well-Being Scale (FACIT-Sp-12) is a brief self-report measure designed to assess the nature and extent of individual's spiritual well-being. This measure (range 0-48), which generates two sub-scales, Faith (the importance of faith/spirituality, range 0-16) and Meaning /Peace (one's sense of meaning and purpose in life, range 0-32). The total score for the FACIT-Sp scale is the sum of the two subscales Faith and Meaning /Peace. It has been demonstrated to have strong internal reliability for both the total score as well as each subscale (coefficient alpha = .87 for the total scale, .88 for the faith factor and .81 for the meaning factor). Higher scores represent a higher level of spiritual well-being, faith or meaning-peace. In addition, strong support for the external validity of this measure has been demonstrated in a several large samples of cancer and AIDS patients and with Spanish speaking populations. Administration time takes approximately 4 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Rosario Costas-Muniz, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (3):
  - MSK at Ralph Lauren, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York
- Ponce Health Sciences University, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org